CLINICAL TRIAL: NCT05738980
Title: Prevention of Postoperative Recurrence of Hepatocellular Carcinoma by Blocking RAK Cells With Anti-TIM-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BJH Biotherapy Center
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-Tim3-blocked RAK cells (Experimental): ubjects were randomly assigned to receive anti-TIM-3 blocked RAK cells or untreated RAK cells.
  Interventions: Biological: Autologous RAK cells
- Unblocked RAK cells (Experimental): ubjects were randomly assigned to receive anti-TIM-3 blocked RAK cells or untreated RAK cells.
  Interventions: Biological: Autologous RAK cells

INTERVENTIONS:
Biological: Autologous RAK cells — Autologous RAK cells were treated by intravenous reinfusion

SUMMARY:
To compare the safety and efficacy of unmodified RAK cells and anti-TIM-3 blocked autologous RAK cells in preventing postoperative recurrence of HCC by postoperative TACE therapy combined with immune cell therapy.

DETAILED DESCRIPTION:
Research process:

Initial screening period (-7 to -1 days)

• Sign an informed consent form;

• Assign screening numbers;

• Assessment of eligibility for initial screening.

1. Day 0 (period 1)

   * Reconfirm the inclusion and exclusion criteria;
   * 50-60ml of anticoagulant peripheral blood was sampled;

   Treatment time:
2. On (±2) days 15 and 16, Autologous RAK cells were reinfused for treatment (cycle 1).
3. TACE was performed on day 28 (±7).
4. Blood drawing from autologous RAK cells in the second cycle (week 10 ±7 days)
5. The second cycle of autologous RAK cell transfusion treatment (12 weeks ±7 days after hepatocellular carcinoma surgery);
6. Blood was drawn from autologous RAK cells in the third cycle (week 22 ±7 days);
7. Reinfusion of autologous RAK cells in the third cycle (week 24 ±7 days);

After completing 3 cycles of treatment, the patients were assessed by the investigator to be under control or remission of disease after treatment, and then they were followed up for treatment

ELIGIBILITY:
Inclusion Criteria:

* 3) Patients diagnosed with HCC by histological examination; 4) According to China Liver Cancer Staging (CNLC) -- Guidelines for the Diagnosis and Treatment of primary liver Cancer of the National Health Commission of the People's Republic of China (2022 edition), patients with stage Ia and stage Ib ⅱA; 5) Undergoing radical resection of HCC; 6) For patients with hepatocellular carcinoma diagnosed by pathology after radical resection, the clinical and pathological characteristics meet one of the following conditions: A. tumor ≥5cm; B. Pathology suggested MVI (microvascular invasion); C. Pathology suggested satellite foci or sub-foci; D. Multiple tumors (number of tumors ≥2); E. AFP & GT; 20 mu g/L; F. Accompanied by hepatic capsule invasion; 7) ECOG score 0 or 1; Child-pugh liver function score A/B (≤7); 8) Neutrophil count ≥1.5×109/L, lymphocyte count ≥1.1×109/L, platelet count ≥80×109/L; Cardiac echocardiography showed that cardiac ejection fraction ≥50%, and 12-lead ECG showed no obvious abnormalities. Oxygen saturation ≥90%; Creatinine clearance rate CG formula ≥50 mL/min; ALT and AST 2.5 x ULN or less; Serum total bilirubin ≤1.5×ULN; 9) The estimated survival time is more than 6 months; 10) Fertile men or women with the possibility of becoming pregnant agree to use effective contraceptive methods (e.g., oral contraceptives, intrauterine devices, controlled sexual desire or barrier contraception combined with spermicide) during the trial and to continue contraception for 3 months after completion of treatment.

Exclusion Criteria:

* 1) Pregnant or lactating women; 2) Previous systemic treatment: cytotoxic chemotherapy drugs within 3 months, targeted drugs within 2 months, interferon and/or interleukin-2 within 3 months, and leukocyte raising drugs within 2 weeks; Have been treated with drugs that target immune regulatory points; 3) Have used immunosuppressive agents (e.g., azathioprine, 6-mercaptopurine, cyclosporine, tisirolimus, everolimus, rapamycin, etc.); Long-term use of corticosteroids; 4) History of thromboembolism within the last 3 months or high risk of pulmonary embolism; 5) Previous use of DC-CIK or CIK cells, autologous RAK/LAK cells or other adoptive immunotherapy; 6) A history of other malignant diseases in the last 5 years (except cured skin cancer and carcinoma in situ of the cervix); 7) Uncontrolled epilepsy, central nervous system diseases, cerebrovascular accidents, or accompanied by other uncontrolled diseases; A history of mental disorders; 8) Clinically severe heart disease (NYHA) grade II or more congestive heart failure or severe arrhythmias requiring medical intervention; 9) Interstitial lung disease ≥2 degrees; 10) Accompanied by fever or infection; 11) Autoimmune diseases, including uncontrolled hypothyroidism and hyperthyroidism; 12) HIV/AIDS or syphilis antibody positive; 13) Allergic to any interferon and interleukin-2 preparations; 14) Participating in other trials within 4 weeks before enrollment; 15) Poor compliance or conditions deemed inappropriate for study inclusion by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
RFS | two years
  Recurrence-free survival (RFS) of postoperative TACE combined with TIM-3 block treated autologous RAK cells to prevent HCC recurrence

SECONDARY OUTCOMES:
OS | 2 years
  Overall survival (OS) of postoperative TACE combined with TIM-3 blocked autologous RAK cells to prevent HCC recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jie Ma, Doctor, Principal Investigator — Beijing Hospital
Locations (1):
- Beijing Hospital Center of Biotherapy, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
After the article was published